CLINICAL TRIAL: NCT02383277
Title: Acute Effects of a Stretching Program of the Rib Cage Muscles on the Regional Distribution of Ventilation and the Diaphragmatic Mobility of Patients With COPD During Exercise: a Randomized Crossover Clinical Trial
Brief Title: Acute Effects of a Stretching Program of the Rib Cage Muscles on Patients With COPD During Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Adriane Borba Cardim, Degree in Physical Therapy, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UFPEFT2015
Record Dates: First submitted 2015-02-13; First posted 2015-03-09 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stretching and Exercise (Experimental): This group undergo a session of stretching aiming flexibility of the rib cage and later at an exercise test with constant load up to the limit of tolerance for exercise bike
  Interventions: Other: Stretching; Other: Exercise
- Control and Exercise (Sham Comparator): This group will carry out the exercise test with constant load up to the limit of tolerance for exercise bike after a period of rest under the same environmental conditions and the experimental group time. During this time the therapist will place their hands but not performing the stretch.
  Interventions: Other: Control; Other: Exercise

INTERVENTIONS:
Other: Stretching — Stretching of the rib cage muscles
  Arms: Stretching and Exercise
Other: Control — Rest without stretching (sham)
  Arms: Control and Exercise
Other: Exercise — Constant load exercise on a bike

SUMMARY:
Investigate the effects of stretching the muscles of the rib cage in individuals with COPD during exercise.

DETAILED DESCRIPTION:
To investigate the effects of a stretching program for the muscles of the rib cage or control in patients with COPD during exercise and / or the immediate post-exercise, using the following parameters:

* Tidal volume (VT), respiratory rate (RR), minute volume (MV), inspiratory time (Tins) and expiratory (T exp).
* Change in volumes of total and regional chest magazines (pulmonary rib cage, abdominal rib cage and abdomen).
* Diaphragmatic mobility.
* electrical muscle activity
* endurance time.
* Dyspnea sensation.

ELIGIBILITY:
Inclusion Criteria:

* Smoking history, occupational or environmental exposure to pollutants and / or symptoms of cough, dyspnea or hypersecretion;
* FEV1 <80% predicted and post-bronchodilator FEV1 / FVC <70% to confirm the diagnosis of airway obstruction not fully reversible bronchodilator therapy;
* Absence of co-morbidities that does not allow the realization of stress (hypertension, severe pulmonary hypertension, myocardial infarction, congestive heart failure, severe dyspnoea);
* Preserved cognitive functioning;
* Sedentary
* Clinically stable during the study period.

Exclusion Criteria:

* Patients with cognitive, hearing or visual deficit;
* Changes in the neuro-musculo-skeletal system which endangers or impairs the assessment;
* Obese
* Not be able to achieve at least three stages of the incremental test.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-10 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Endurance tolerance as measured by the duration of the exercise | Participants will be followed for the duration of the exercise, an expected average of 10 minutes
Dyspnea as measured by Borg Escale | Participants will be followed for the duration of the exercise, an expected average of 10 minutes

SECONDARY OUTCOMES:
Diaphragm mobility measured by ultrasound | Participants will be followed for the duration of the stretching and the exercise, an expected average of 60 minutes
Volumes of the chest wall measured by pletismography optoelectronic | Participants will be followed for the duration of the stretching and the exercise, an expected average of 60 minutes
Muscle electrical activity measured by surface electromyography | Participants will be followed for the duration of the stretching and the exercise, an expected average of 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Adriane Cardim, Graduated, Principal Investigator — Universidade Federal de Pernambuco